CLINICAL TRIAL: NCT06671444
Title: A Phase 1 Open-Label Single-Dose Study to Assess the Pharmacokinetics and Safety of YZJ-1139 in Subjects With Severe Renal Impairment and Renal Impairment
Brief Title: Pharmacokinetics and Safety Study of YZJ-1139 in Subjects With Severe Renal Impairment and Normal Renal Impairment
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Haiyan Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YZJ-1139-1-12
Record Dates: First submitted 2024-10-31; First posted 2024-11-04 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Insomnia; Renal Impairment
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Renal Insufficiency

STUDY DESIGN:
Intervention Model Description: single dose
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Severe Renal Impairment (Experimental)
  Interventions: Drug: YZJ-1139
- Group B: Normal Renal Impairment (Experimental)
  Interventions: Drug: YZJ-1139

INTERVENTIONS:
Drug: YZJ-1139 — Single oral dose, 20 mg tablet

SUMMARY:
Objective：

1. To evaluate the pharmacokinetics of YZJ-1139 tablets in patients with severe renal impairment and in subjects with normal renal impairment.
2. To evaluate the safety of YZJ-1139 tablets in patients with severe renal impairment and in subjects with normal renal impairment.

ELIGIBILITY:
Entry criteria（Group A-Severe Renal Impairment Group）:

1. Male or female subjects aged 18-65 years (inclusive).
2. Weight ≥ 50.0 kg for males, or ≥ 45.0 kg for females, and body mass index (BMI) in the range of 19.0 ~ 28.0 kg/m2 (inclusive).
3. Subjects has been diagnosed with chronic kidney disease (more than 3 months) and have stable renal function (absolute eGFR change within 25% at least 1 month at screening), absolute eGFR at screening meets the renal function classification criteria, severe renal insufficiency: 15 ~ 29 mL/min;.
4. Subjects of childbearing potential (including partners) have no family planning or donate sperm/eggs from 2 weeks before screening to 3 months after dosing, and voluntarily take appropriate contraceptive measures;
5. Subjects who are able to understand and willing to complete the study in strict compliance with the clinical protocol and sign the informed consent form

Exclusion criteria(Group A-Severe Renal Impairment Group):

1. Allergic constitution, such as those with a known history of allergies to drugs, food or other substances, or those with a history of allergies to YZJ-1139 tablets or similar orexin receptor antagonist drugs and excipients;
2. Subjects with difficulty swallowing tablets, and special dietary requirements who cannot accept a unified diet;
3. Subjects who have poor peripheral venous access or cannot tolerate venous puncture or have a history of needle and blood fainting;
4. Subjects who have undergone surgery within 30 days prior to screening, or plan to undergo surgery during the study;
5. Individuals with a history of paroxysmal sleep disorder, obstructive sleep apnea, complex sleep behavior (such as dream walking, driving in dreams, etc.), severe unconscious hypoglycemia, stroke, epilepsy, and other psychiatric disorders (including anxiety, depression, etc.), convulsive diseases, and sudden onset of illness;
6. Patients who have received kidney transplantation and/or require renal dialysis during the trial.
7. Except for the disease causing renal dysfunction itself, those who have previously or currently suffered from other serious systemic organ diseases, including respiratory, digestive, endocrine, malignant tumor, blood, mental/nervous system serious diseases, which were judged by the investigator to be unsuitable for participation in this trial;
8. Subjects with ALT and/or AST > 2 ULN and/or TBIL > 1.5 ULN, Hb < 80 g/L, QTcF > 450 ms in males and QTcF > 470 ms in females by ECG.
9. Subjects with poorly controlled hypertension (systolic blood pressure ≥ 160 mmHg and/or diastolic blood pressure ≥ 100 mmHg) or heart rate > 120bmp.
10. Patients with diabetic nephropathy HbAlc (glycosylated hemoglobin) > 8.5% or fasting blood glucose > 8.5 mmol/L, or stable treatment regimen for less than 1 month before screening.
11. Subjects with active HBV infection (HBV DNA copy number ≥ 104 copies/mL must be excluded if HBsAg is positive), or those who are positive in any index screening of HCV, human immunodeficiency virus antibody, syphilis antibody.
12. Subjects with a history of drug abuse, drug use within 6 months before screening, or positive drug abuse screening;
13. Subjects who frequently consume alcohol within 3 months prior to screening, i.e., consuming more than 14 units of alcohol per week (1 unit = 360 mL of beer or 45 mL of 40% spirits, or 150 mL of wine), or who cannot stop using any alcohol products during the study, or alcohol breath test result > 0.0 mg/100 mL;
14. Subjects who have donated blood or experienced massive blood loss (> 400 mL) within 3 months prior to screening, received blood transfusions or used blood products, planned to donate blood during the trial period or within 1 month after the end of the trial;
15. Subjects who have consumed excessive tea, coffee and/or caffeine-containing beverages (more than 8 cups, 1 cup ≈ 250 mL) daily during the 3 months before screening;
16. Subjects smoke an average of 5 or more cigarettes per day within 3 months prior to screening, or those who cannot stop using any tobacco products during the study;
17. Subjects who have participated in any clinical trial and have used clinical trial drugs within 3 months prior to screening, or plan to participate in other clinical trials during the study;
18. Subjects who have received vaccination within 30 days prior to screening, or plan to receive vaccination during the study;
19. Subjects who have used any CYP3A4 enzyme inducer or inhibitor within 30 days (or 5 half-lives, whichever is longer) prior to administration;
20. Subjects who have used any prescription drugs, over-the-counter drugs, vitamin products, health products or Chinese herbal medicines other than those for the treatment of renal insufficiency and or its concomitant chronic diseases within 14 days before administration;
21. Subjects who started taking new drugs, dosage forms or adjusted current doses for the treatment of chronic kidney disease and its combined chronic diseases within 14 days before administration;
22. Subjects who have consumed special diets (including grapefruit, chocolate, xanthine-rich or alcohol-rich foods/beverages) within 48 h before administration;
23. Lactating women, or women who test positive for pregnancy;
24. Subjects with acute illness from screening to prior to administration;
25. Those who, in the opinion of the investigator, are not suitable for inclusion.

Entry criteria（Group B-Healthy Subject Group）:

1. Subjects aged 18 to 65 years (inclusive), matched with renal impairment for age and sex (each subject in Group B within± 10 years of the mean for Group A and with a mean of ± 1 case for Group A by gender)；
2. Weight ≥ 50.0 kg for males, or ≥ 45.0 kg for females, and body mass index (BMI) in the range of 19.0 ~ 28.0 kg/m2 (inclusive), matched to BMI with renal impairment group (each subject in Group B within ±15% of mean in Group A by BMI).
3. Normal renal function, 90 mL/min ≤ absolute eGFR < 130 mL/min;
4. Subjects with normal physical examination, vital signs (normal range refers to central SOP), 12-lead ECG, laboratory tests, imaging and abdominal ultrasonography results during the screening period or abnormal but no clinical significance as judged by the investigator;
5. Subjects of childbearing potential (including partners) have no family planning or donate sperm/eggs from 2 weeks before screening to 3 months after dosing, and voluntarily take appropriate contraceptive measures;
6. Subjects who are able to understand and willing to complete the study in strict compliance with the clinical protocol and sign the informed consent form.

Exclusion criteria(Group B-Healthy Subject Group):

1. Allergic constitution, such as those with a known history of allergies to drugs, food or other substances, or those with a history of allergies to YZJ-1139 tablets or similar orexin receptor antagonist drugs and excipients;
2. Subjects with difficulty swallowing tablets, and special dietary requirements who cannot accept a unified diet;
3. Subjects who have poor peripheral venous access or cannot tolerate venous puncture or have a history of needle and blood fainting;
4. Individuals with a history of paroxysmal sleep disorder, obstructive sleep apnea, complex sleep behavior (such as dream walking, driving in dreams, etc.), severe unconscious hypoglycemia, stroke, epilepsy, and other psychiatric disorders (including anxiety, depression, etc.), convulsive diseases, and sudden onset of illness;
5. Subjects who have a history of other serious diseases and chronic diseases such as respiratory system, circulatory system, digestive system, urinary system, blood system, endocrine system, immune system, nervous system, mental system;
6. Those who are positive in any index screening of hepatitis B virus surface antigen, Treponema pallidum-specific antibody, human immunodeficiency virus antibody,or hepatitis C virus antibody；
7. 12) Subjects with a history of drug abuse, drug use within 6 months before screening, or positive drug abuse screening;
8. Subjects who frequently consume alcohol within 3 months prior to screening, i.e., consuming more than 14 units of alcohol per week (1 unit = 360 mL of beer or 45 mL of 40% spirits, alcohol or 150 mL of wine), or who cannot stop using any alcohol products during the study, or whose alcohol breath test result > 0.0 mg/100 mL;
9. Subjects who have donated blood or experienced massive blood loss (> 400 mL) within 3 months prior to screening, received blood transfusions or used blood products, planned to donate blood during the trial period or within 1 month after the end of the trial;
10. Subjects who have consumed excessive tea, coffee and/or caffeine-containing beverages (more than 8 cups, 1 cup ≈ 250 mL) daily during the 3 months before screening;
11. Subjects smoke an average of 5 or more cigarettes per day within 3 months prior to screening, or those who cannot stop using any tobacco products during the study;
12. Subjects who have participated in any clinical trial and have used clinical trial drugs within 3 months prior to screening, or plan to participate in other clinical trials during the study;
13. Subjects who have undergone surgery within 30 days prior to screening, or plan to undergo surgery during the study;
14. Subjects who have received vaccination within 30 days prior to screening, or plan to receive vaccination during the study;
15. Subjects who have used any CYP3A4 enzyme inducer or inhibitor within 30 days (or 5 half-lives, whichever is longer) prior to administration;
16. Subjects who have taken any prescription drugs, over-the-counter drugs, health products, vitamins, and Chinese herbal medicines within 14 days before administration;
17. Subjects who have consumed special diets (including grapefruit, chocolate, xanthine-rich or alcohol-rich foods/beverages) within 48 h before administration;
18. Lactating women, or women who test positive for pregnancy;
19. Subjects with acute illness from screening period to pre-dose;
20. Those who, in the opinion of the investigator, are not suitable for inclusion.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2024-06-03 (Actual); Primary Completion 2024-11-10 (Estimated); Study Completion 2024-12-25 (Estimated)

PRIMARY OUTCOMES:
Area Under the Plasma Concentration-time Curve From Time 0 to the Last Measurable Concentration (AUC0-t) of YZJ-1139 | From Day 1 to Day 3
  AUClast is defined as the concentration of drug from time zero to the last observable concentration
Area Under the Plasma Concentration-time Curve From Time 0 Extrapolated to Infinity (AUC0-∞) of YZJ-1139 | From Day 1 to Day 3
  AUCinf is defined as the concentration of drug extrapolated to infinite time
Maximum Observed Plasma Concentration (Cmax) of YZJ-1139 | From Day 1 to Day 3
  Cmax is defined as the maximum concentration of drug
Apparent Oral Clearance (CL/F) of Entrectinib | From Day 1 to Day 3
  CL/F is defined as the apparent oral clearance following administration of the drug
The Apparent Volume of Distribution (Vz/F) of Entrectinib | From Day 1 to Day 3
  Vz/F is defined as the apparent volume of distribution of the drug
Time of Maximum Observed Plasma Concentration (Tmax) of Entrectinib | From Day 1 to Day 3
  Tmax is defined as the time (observed time point) of Cmax
Apparent Terminal Elimination Half-life (t1/2) of Entrectinib | From Day 1 to Day 3
Mean Residence Time (MRT0-t) of YZJ-1139 | From Day 1 to Day 3
Renal Excretion (Ae) of YZJ-1139 | From Day 1 to Day 3
renal clearance (CLR) of YZJ-1139 | From Day 1 to Day 3
Percentage of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | From Day 1 to Day 7

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Zhongda Hospital Southeast University, Nanjing, Jiangsu
  - The First Affiliated Hospital of Bengbu Medical University, Bengbu
  - The First Affiliated Hospital of Xuzhou Medical University, Xuzhou